CLINICAL TRIAL: NCT06724003
Title: The Effect of Computer-based Virtual Reality Simulation on Nursing Students' Knowledge, Self-confidence and Satisfaction Levels: Oral Care Practice in Unconscious Patient
Brief Title: The Effect of Simulation on Nursing Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Giresun University (Other)
Responsible Party: Principal Investigator, AsumanCobanoglu, Assistant Professor, Giresun University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: GiresunU-SBF-AC-01
Record Dates: First submitted 2024-11-26; First posted 2024-12-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Nursing Student
Keywords: virtual reality; nursing student; confidence; satisfaction; simulation
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This study is a randomized controlled experimental trial.
Who Masked: Outcomes Assessor
Masking Description: Statistical analyses and data reporting of the study will be carried out by statistical experts who are not among the researchers and are not familiar with the research application. The study was blinded in terms of outcome measures, statistical analysis and reporting to prevent statistical and reporting bias. In this context, the statistical expert was blinded; the researchers and students were not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Computer-based simulation of virtual reality . (Experimental): Interactive virtual reality simulation group will practice oral care in the unconscious patient with interactive virtual reality simulation after the oral care practice in the unconscious patient is demonstrated on a low reality patient manikin. After the application, a briefing will be given to the participants and the application will be discussed in detail. Participants will perform oral care in the unconscious patient on a low-reality patient manikin 15 days after the simulation application.
  Interventions: Other: Computer-based virtual reality simulation
- Low-reality patient model group (No Intervention): Participants will be demonstrated the unconscious patient oral care practice with a low-reality patient manikin by the researcher nurse faculty member. Participants will perform the application on the low-reality patient manikin. After the application, participants will be briefed and talked about the application. Oral care of the unconscious patient will be practiced on a low-reality patient manikin 15 days after the application.

INTERVENTIONS:
Other: Computer-based virtual reality simulation — The computer-based virtual practice simulation was created as a single scenario for oral care practice in the unconscious patient. The scenario software was created and designed by the researcher who is an IT specialist. In the formation phase of the scenario, the software was realized by working together with the researcher, the expert faculty member, the nurse and the informatics specialist for the photographs required for the virtual reality application and the steps of the scenario software.
  Other Names: Experimental group
  Arms: Computer-based simulation of virtual reality .

SUMMARY:
The aim of this study was to evaluate the effect of computer-based virtual reality (VR) simulation on students' knowledge, satisfaction and self-confidence in teaching oral care practice in the unconscious patient.

Oral care practice in the unconscious patient is one of the important nursing interventions in terms of patient health, which is given from the first years of nursing education.

This study is a randomized controlled experimental research. The study will be conducted with first-year nursing students enrolled in a university in Turkey. The sample of the study will consist of 68 nursing students. The data will be collected by Student Information Form, Oral Care Practice Information Form, Student Satisfaction in Learning and Self-Confidence Scale.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the effect of computer-based virtual reality (VR) simulation on students' knowledge, satisfaction and self-confidence in teaching oral care practices in the unconscious patient.

Oral care practice in the unconscious patient is one of the important nursing interventions in terms of patient health, which is given from the first years of nursing education.

This study is a randomized controlled experimental research. The study will be conducted with first year nursing students enrolled in a university in Turkey. The sample of the study will consist of 68 nursing students. Participants will be randomized into a computer-based virtual reality simulation group (n=34) and a low-reality patient manikin group (n=34). The research data will be collected by Student Information Form, Oral Care Practice Information Form, Student Satisfaction in Learning and Self-Confidence Scale.

Participants in the experimental and control groups will be informed about the methodology, aims and objectives of the study and their consent to participate in the study will be obtained both verbally and in writing. The theoretical content of the course will be given to the participants by the researcher faculty member using power point presentation and question-answer method. After the theoretical training, students will fill in the Student Information Form and Oral Care Practice Information Form.

After the forms are filled in, the students in both groups will be taken to the laboratory where the low-reality patient model is located. Students will be given a checklist showing the steps of oral care practice in the unconscious patient before the application. Oral care application steps in the unconscious patient will be shown to the students on the low-reality patient model by the researcher nurse faculty member. The participants in the control group will perform the oral care skill in the unconscious patient on the model.

The participants in the experimental group will then be taken by the researchers to the laboratory where the computer-based interactive VR simulation is used. Participants will be given a checklist showing the oral care application steps in the unconscious patient before the simulation application. Participants will be given preliminary information about the computer-based interactive VR simulation system and its application. Oral care practice in the unconscious patient will be demonstrated to the participants in the interactive VR simulation by the research nurse faculty member. Participants will be allowed to ask questions during the simulation and their questions will be answered. After the hands-on training, the participants will be taken to the laboratory one by one to practice oral care in the unconscious patient with the interactive VR simulation. While the participant is practicing oral care in the unconscious patient in the simulation application, the researcher faculty member will control the oral care practice of the participants. While the participant is practicing oral care in the unconscious patient in the simulation application, the researcher faculty member will check the skill steps on the participants' oral care practice checklist.

After a participant finishes the practice and leaves the laboratory, another participant will be called to the room for the practice and each participant will be given an average of 10 minutes for the practice. After the application is completed, each participant will fill in the Oral Care Application Information Form and the Student Satisfaction and Confidence in Learning Scale. After the implementation process, information sessions will be held with the participants in the experimental and control groups. These sessions will be held with groups of 5-6 students. Reassuring and open communication was established with the participants and they were encouraged to think. In the debriefing session, the participants will be asked "What did you do well?" and "What would you do differently if you had the opportunity to experience this simulation again?" and will be asked to give reflective answers. Participants will be given feedback about their performance by the trainer in line with the skill checklists used. Participants in the experimental and cortol groups will be asked to practice oral care in the unconscious patient in the simulation and low-reality patient mannequin 15 days after the oral care practice in the low-reality patient mannequin in the unconscious patient. Participants will fill in the Oral Care Practice Information Form and the Student Satisfaction and Self-confidence in Learning Scale after completing the practices.

ELIGIBILITY:
Inclusion Criteria:

* Basic Principles and Concepts in Nursing course for the first time,
* Volunteering to participate in the study.

Exclusion Criteria:

* Graduating from a health-related high school or an associate's or bachelor's degree from a health-related university,
* Having received training on oral care practice in the unconscious patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-02-25 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Student Satisfaction and Self-confidence in Learning Scale (SCLS) | two weeks
  The scale developed by Jeffries & Rizzolo consists of 13 items. The Turkish validity and reliability study of the scale was conducted by Ünver et al. In this form, the number of items was reduced to 12. There are 5 items in the "Satisfaction with Current Learning" subscale and 7 items in the "Confidence in Learning" subscale. The Cronbach alpha value in the Turkish version is 0.85 for satisfaction with learning and 0.77 for self-confidence in learning. The scale is a 5-point Likert scale; responses are measured with values between 1 (strongly disagree) and 5 (strongly agree). Scale scores are obtained by dividing the sum of the sub-dimensions by the number of items. Accordingly, the minimum score is 1 and the maximum score is 5. It is thought that the higher the score obtained from the scale, the higher the satisfaction and self-confidence.

SECONDARY OUTCOMES:
Student Information Form | two weeks
  It was prepared by the researchers based on previous studies in the literature. The form consists of 9 questions inquiring the demographic and academic information and technology usage characteristics of the participating students (gender, year of birth, academic average, computer use, etc.).
Oral Care Practice Information Form | two weeks
  This form was developed by the researchers by reviewing the relevant literature in accordance with the oral care application steps in unconscious patients. After the relevant form was developed by the nurse faculty member, it was also examined and edited by 2 nurse faculty members who are experts in the field. The form includes 18 items for oral care practice in unconscious patients. The statements in the form consist of 3 options as true, false and don't know/no idea. In the form, the "Correct" response of the students to the statements corresponds to 1 point, and "Incorrect" or "Don't Know/No Idea" responses correspond to 0 points. Students can get a maximum of 18 points and a minimum of 0 points from this form.

CONTACTS AND LOCATIONS:
Overall Officials: Asuman Çobanoğlu Assistant Professor, PhD., Study Chair — Giresun University Faculty of Health Sciences
Locations (1):
- Giresun University Faculty of Health Sciences, Giresun, Piraziz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
It will be shared when requested from the researcher.